CLINICAL TRIAL: NCT00672308
Title: Efficacy of Benefiber-Added, Reduced-Osmolarity WHO-ORS in the Treatment of Cholera in Adults
Acronym: ORS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Collaborators: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002-034
Record Dates: First submitted 2008-05-03; First posted 2008-05-06 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2004-12

CONDITIONS: Cholera
Keywords: Cholera, benefiber, ORS
MeSH Terms: conditions — Cholera; Osteoarthritis | interventions — ORALIT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Benefiber (25 g/L)
  Interventions: Other: Benefiber with ORS; Other: the reduced-osmolarity WHO-ORS without added Benefiber
- 2 (Experimental): Benefiber (50 g/L)
  Interventions: Other: Benefiber; Other: Benefiber with ORS
- 3 (Experimental): the reduced-osmolarity WHO-ORS without Benefiber.
  Interventions: Other: Benefiber with ORS; Other: the reduced-osmolarity WHO-ORS without added Benefiber

INTERVENTIONS:
Other: Benefiber
  Arms: 2
Other: Benefiber with ORS — Benefiber (50 g/L)-supplemented, reduced-osmolarity WHO-ORS
  Arms: 3
Other: Benefiber with ORS
  Arms: 1
Other: Benefiber with ORS
  Arms: 2
Other: the reduced-osmolarity WHO-ORS without added Benefiber
  Arms: 1
Other: the reduced-osmolarity WHO-ORS without added Benefiber
  Arms: 3

SUMMARY:
In cholera, the function of small intestine is affected resulting in increased secretion of electrolytes and water and their reduced absorption leading to profuse watery diarrhoea. The human colon has the capacity to absorb water and electrolytes. A number of recent studies have shown that short chain fatty acids (SCFAs) such as acetate, butyrate and propionate stimulates absorption of sodium in the colon, which is not affected by cyclic AMP. It has also been shown that SCFAs inhibits c-AMP mediated chloride secretion in the colon. Benefiber (partially hydrolyzed guar gum) is water soluble fibre, and when added to ORS it undergoes fermentation in the colon liberating SCFAs. SCFAs not only serves as metabolic fuel to the enterocytes but they also enhance colonic absorption of salts and water. Thus, they have potentials to reduce the severity of diarrhoea in patients with cholera. The aim of this study is to assess the efficacy of Benefiber-added WHO-ORS in the management of adults with cholera. In this randomized, controlled clinical trial, a total of 174 adult males with cholera would be studied. Study patients would be selected from those who attend the Dhaka Hospital of ICDDR,B with a history of diarrhoea of less than 24 hours and signs of severe dehydration. They would be rehydrated using intravenous fluid (cholera saline) over 4 hrs during which a stool specimen would be subjected for dark-field microscopy for identification of V. cholerae. Those identified to have cholera would be randomized in equal numbers to receive either: a) Benefiber (25 g/L) added WHO-ORS, b) Benefiber (50 g/L) added to the new formulation (Na+ 75, glucose 75, Cl- 65, K+ 20 mmol/L, citrate 10 mmol/L, osmolarity 245 mosmol/L) of WHO-ORS , or c) the same WHO-ORS but without Benefiber for maintenance of hydration until resolution of diarrhoea. All patients would be treated with a single, 300 mg dose of doxycycline capsules and would be provided with the standard hospital diets. Fluid intake (intravenous fluid, ORS, and plain water) and output (stool, urine, and vomit) will be measured for each 6-hourly periods of the study. Patients would be hospitalized until resolution of their diarrhoea. Stool output, intake of intravenous fluid and ORS, the duration of diarrhoea, and the proportion of patients requiring "unscheduled intravenous fluid therapy" would be compared between the treatment groups. If Benefiber is found effective, it would be possible to formulate improved ORS for better case management of cholera.

DETAILED DESCRIPTION:
Considerable interest has recently been generated on dietary fibers (DF), and soluble fibers have emerged both as a subject for research and therapeutic applications. The 'fiber hypothesis', put forward by Denis Bukitt and Hugh Trowel (1-4), suggests that consumption of unrefined carbohydrate food protects against many western ailments including colon cancer, diverticular disease, appendicitis, constipation, haemorrhoids, diabetes, heart disease, gall stones, and obesity among others. In the line of this hypothesis, many basic laboratory and clinical works have been done. The term 'dietary fiber' has been used to denote plant polysaccharides and lignin that are resistant to hydrolysis by human digestive enzymes (5,6). The detailed chemistry and metabolism of DF have also been studied (7-10). The classification of fiber is based on their chemical structures (11), and they can be divided into non-polysaccharides and non-starch polysaccharides. Lignin is the only non-polysaccharide fiber, which is a polymer of phenolic alcohol that is water insoluble. The non-starch polysaccharide can be divided into cellulose and non-cellulose fiber. Cellulose consists of un-branched D-glucose chains in 1,4-ß linkage and is water insoluble. Non-cellulose polysaccharides include hemicelluloses, mucillages, gums and pectins, and they consists of various ß linkages of wide variety of hexose and pentose sugars. The polysaccharide chains are heteroglycans (chains with more than one type of monosaccharide). The hemicellulosic materials are polymers of xylose, mannose and glucose with side chains of galactose and arabinose. The pectic substances are polymers of galacturonic acids. Likewise, the gums and mucillages are branched carbohydrate polymers (e.g. gum, which is a linear mannan with galactose side chains). Non-cellulose polysaccharides vary in degree of their water solubilities (7,9,10).

In man, fiber is mainly degraded in the large intestine by the bacterial flora. Many of the effects of fiber on stool output arise from this degradation. The main products of fiber fermentation are short chain fatty acids (SCFAs) including acetate, propionate and butyrate, which are the major anions in the colon. Bacteria utilize SCFAs and proliferate, absorbing water from the colonic epithelium in the course of their metabolism, and thus decrease the free water content in the lumen (11). The SCFAs that are not utilized by the bacteria are largely absorbed by the colon (12). Their transepithelial transport is associated with stimulation of sodium transport from the colon in several species including human (13-15). This effect may be particularly important in acute diarrhoeal diseases where purging, and associated reduced food intake might deplete the colon of SCFAs leading to colonic dysfunction (16, 17). Thus, luminal SCFAs levels in the colon might influence the clinical course of acute diarrhoeal diseases. SCFAs have also been shown to be clinically important in one diarrhoeal disease in animal -transmissible gastroenteritis of swine (18). Animals infected with the virus develop acute enteritis with marked fluid loss from the small intestine. Young animals develop severe diarrhoea as their colonic mucosa is incapable of absorbing fluid, whereas older infected animals has been shown to have increased colonic absorption by about six-folds over the controls. This compensatory response prevents severe diarrhoea and is related to the development of colonic fermentation with the production of SCFAs.

Cholera is a disease of humans affecting the small intestine where fluid and electrolyte secretion is increased while their absorptions are decreased leading to profuse watery diarrhoea. As the human colon has the capacity to absorb water and electrolyte (19), some compensation is expected reducing the diarrhoeal loss. In recent studies (20, 21) SCFAs have been shown to stimulate sodium absorption in the colon, an effect that is not influenced by c-AMP, and additionally they have been found to inhibit cyclic AMP-mediated chloride secretion in the colon.

The SCFA-enhanced colonic absorption of water and electrolytes might be exploited in the treatment of acute diarrhoeal diseases. Oral rehydration therapy has dramatically changed the management of acute diarrhoeal disease. Yet, oral rehydration therapy is in the process of being improved. Cereal-based oral rehydration solutions (ORS) have been shown to reduce the stool volume by about 30% to 40% compared to the WHO-ORS (22, 23). It is possible that, at least a part of their effect on stool volume reduction might be attributed to SCFAs produced by unabsorbed carbohydrate including dietary fiber in the colon. Diversion colitis is an inflammatory process affecting the bypassed colon and rectum following surgical diversion of faecal stream (24). The inflammation disappears after surgical re-anastomosis, where topical steroids are usually ineffective (25). Rectal instillation of SCFAs has resulted in the disappearance of symptoms and endoscopic change over a period of 4-6 weeks; remission has been maintained for over a year by regular rectal SCFAs treatment (26). These findings suggest that SCFAs also play a role in mucosal healing in colitis

The colonic epithelial cells utilize SCFAs as source of energy for their various metabolic activities (27, 28). Human colonocytes use butyrate in preference to glucose, glutamine or ketone bodies as fuel source (27). Thus, in contrast to small intestinal cells, colonic epithelial cells derive the major part of their energy supply from the lumen rather than from the blood. Depriving luminal nutrition of the mucosa has been found to induce fluid secretion (29). The lack of luminal SCFAs in the colon may be involved in special diarrhoeal states such as diversion colitis and antibiotic associated diarrhoea. Diarrhoea is not uncommon after abdominal operations, particularly after closure of a temporary colostomy (30). Although there is no proof, this postoperative diarrhoea might be attributed to lack SCFAs in the colon, which might perhaps be reversed by the intake of fermentable fiber (31). Lengthy preoperative bowel preparation by antibiotic and lavage, and diminished oral nutrition probably contributes to postoperative diarrhoea. Lack of luminal SCFAs can similarly explain the diarrhoea often seen in the terminal stages of malnutrition and starvation. In these conditions, intestinal infections might not always be implicated and it seems likely that diarrhoea is a manifestation of organ-specific malnutrition of the colon (32). Diarrhoea is often associated with the use of broad-spectrum antibiotics, and colonization by toxin producing clostridium difficile accounts for only a third of these cases (33). The use of antibiotics suppresses the formation of SCFAs from fermentable carbohydrate (34), a feature that might also be responsible for diarrhoea. Although there are lots of data suggesting antidiarrhoeal effect of fermentable fibers, their therapeutic application in diarrhoeal disease is yet to be examined. Some recent clinical studies have demonstrated the beneficial effect of dietary fiber in treatment of adult cholera (35) and in the treatment of children with acute diarrhoea (36). In children with acute diarrhoea, Benefiber-added ORS has been observed to reduce the mean duration of diarrhoea by 16 hours, (74 vs. 90 h; p <0.05). Further studies are required to evaluate the effect of Benefiber in reducing severity and duration of cholera, a form of severe dehydrating diarrhoea.

Guar gum: a soluble fiber

Guar gum is a dietary fiber obtained from the endosperm of the seeds of the Indian cluster bean (Cyanopsis tetragonolobus) of the family Leguminosae. The guar plant is a pod bearing, nitrogen-fixing legume, which has been grown for centuries in India and Pakistan, where it is one of the principal crops and is used as food for both humans and animals. It is now being grown in America for use in various industries (food, cosmetic and paper industries) (37).

Chemically, guar gum is a non-starch polysaccharide, a galactomannan, which on contact with water form a highly viscous gel. In the colon, guar gum is fermented to form SCFAs. Initially, guar gum was used as thickener and emulsion stabilizer in food processing on the basis of its gelling property (37). Our present interest about guar gum is its therapeutic use as a dietary fiber.

"Benefiber" (partially hydrolyzed guar gum)

Guar gum forms gel with water, is rather viscous, and thus unsuitable for therapeutic uses (e.g. in liquid enteral nutrition). Benefiber is a partially-hydrolized (in vitro by the enzyme endo-B-mannase) guar gum, which is a soluble fiber. It is expected that Benefiber will be readily utilized by colonic microflora with the production of the same products of fermentation as the guar gum. The partial hydrolysis of the guar gum (e.g. Benefiber) results in significant reduction in the viscosity of the solution. It is also expected that it will not cause any delay in gastric emptying and also will not interfere with normal absorption of macronutrients (carbohydrate, protein and fat). In one study (38), the addition of Benefiber to a liquid formulation of diet significantly delayed the colonic transit time without affecting the oro-caecal transit time. The result of another recent study (39) in Liestal, Switzerland observed that the Benefiber did not affect the absorption of glucose, amino acid and fat.

Benefiber was chosen for this study for several reasons. First, it is partially-hydrolyzed guar gum (PHGG), and it completely dissolves in water making a clear solution. Second, other fibers are usually viscous, and thus not suitable for use in ORS; the amylase-resistant starch is not soluble and it only makes a suspension. Third, in in vitro studies of fermentation, using fresh faecal inoculate, SCFAs production was observed to be highest with PHGG in comparison with the other commercial fiber substitutes (40). Fourth, in our study in non-cholera diarrhoea in children, we observed PHGG to be clinically useful (36). In this study (36), we used PHGG in a dose of 20g/L. This dose was selected arbitrarily on the basis of standard dose used in the preparation of liquid formulation diets. In the proposed study, we would like to test two different doses (25 g/L and 50 g/L) to determine if there is an additional benefit of increasing the dose.

Based on the findings of our previous study as well as studies done elsewhere, we are very hopeful that the addition of Benefiber to WHO-ORS would lead to its fermentation in the colon resulting in the production of SCFAs, which would improve colonic function including colonic absorption of salt and water and thus reduce the stool output as well as shorten the duration of diarrhoea in adults with cholera.

Safety issue of Benefiber

Benefiber is a food material obtained from vegetable source has been used in cereals, juices, shakes, yogurt, soups, backed goods, and as a fiber source in enteral nutrition products. It has undergone extensive toxicity testing and found to be safe (41). In human volunteer studies (38, 39), enteral nutrition products supplemented with Benefiber 20 g/L found to be safe. Two clinical trials (36, Alam et al., unpublished data) in children have been performed in ICDDR,B recently - in one study ORS was supplemented with Brenefiber 20 g/L and in other study comminuted chicken-based diet was supplemented with Benefiber 20 g/L. No adverse effects have been noted in these studies. In the proposed study, Benefiber will be supplemented with ORS either 25 g/L or 50 g/L for the treatment of adult cholera. As the cholera patients have profuse watery stools with short transit time, 50% of fibers are expected to excrete through stool unchanged. As the treatment of cholera is for a short duration (2-3 days), so we do not anticipate any adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Age: 15 - 55 years
* Gender: Male (women would be excluded due to difficulties in separation of their urine from stools, particularly in those with severely dehydrated and associated mental obtundation).
* Duration of diarrhoea: 24 hours or less
* Clinical signs and symptoms of severe dehydration.
* Demonstration of V. cholerae in dark-field microscopy of a fresh stool specimen
* Written informed consent for participation in the study (for patients with temporary inability to provide consent due to their severe dehydration and mental obtundation, initial consent would be obtained from their attendants; however, the consent process would be re-applied to the patients when they are fully oriented)

Exclusion Criteria:

* Chronic or iatrogenic diarrhoea
* Dysentery (presence of visible blood in stool)
* History of receiving antimicrobial or antidiarrhoeal drugs prior to admission
* Presence of concomitant infection or underlying disease, which might complicate diagnosis and/or assessment of response to study interventions
* History of renal or hepatic dysfunction
* Failure to obtain informed consent

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2003-05; Primary Completion 2005-02 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
total and 24-hourly watery stool output | 24 months

SECONDARY OUTCOMES:
ORS intake and duration of diarrhoea, Clinical success (and failure), success (and failure) of oral rehydration therapy, and the proportion of patients requiring "unscheduled intravenous fluid therapy" | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- ICDDR,B, Dhaka, Bangladesh

REFERENCES:
- [Derived] Alam NH, Ashraf H, Sarker SA, Olesen M, Troup J, Salam MA, Gyr N, Meier R. Efficacy of partially hydrolyzed guar gum-added oral rehydration solution in the treatment of severe cholera in adults. Digestion. 2008;78(1):24-9. doi: 10.1159/000152844. Epub 2008 Sep 4. PMID 18769066